CLINICAL TRIAL: NCT07298733
Title: The Value of Interleukin-1β and Interleukin-33 Genetic Expression in the Pathogenesis and Differentiation of Primary ITP and SLE-Related Thrombocytopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, Assistant professor, Sohag University
Other Study IDs: Soh-Med-25-10-10PD
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia; System; Lupus Erythematosus
Keywords: gene expression; ITP; inflammation; autoimmune
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Lupus Erythematosus, Systemic; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — • 5 ml venous peripheral blood collected under sterile conditions.
  Separation of PBMCs (peripheral blood mononuclear cells).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Systemic lupus erythematosis: patients proved with SLE
  Interventions: Diagnostic Test: measuring gene expression
- Idiopathic thrombocytopenic purpura: patients proved with ITP
  Interventions: Diagnostic Test: measuring gene expression
- Normal controls: normal persons showing no disease matching age and gender
  Interventions: Diagnostic Test: measuring gene expression

INTERVENTIONS:
Diagnostic Test: measuring gene expression — * 5 ml peripheral blood collected under sterile conditions.
  * Separation of PBMCs (peripheral blood mononuclear cells). for :
    1. RNA Extraction: from PBMCs.
    2. cDNA Synthesis: using reverse transcriptase.
    3. Gene Expression Analysis using Quantitative Real-Time PCR (qRT-PCR)

SUMMARY:
Primary immune thrombocytopenia (ITP) is an autoimmune- mediated acquired bleeding disorder, defined as a platelet count less than 100×109/L without other causes of isolated thrombocytopenia. The etiology of ITP is complex and heterogeneous, and as no specific biomarkers are indicating its presence, ITP remains a diagnosis of exclusion. The heterogeneous nature of ITP is evident in the differences in clinical presentation and response to regular treatment among patients and the multiple mechanisms that have been forwarded to account for it, such as autoantibodies, T cell dysregulation, and impaired megakaryocytes. Except primary ITP, all forms of immune-mediated thrombocytopenia is defined as secondary ITP. Secondary ITP has several causes, including autoimmune diseases such as systemic lupus erythematosus

DETAILED DESCRIPTION:
SLE is a complex autoimmune disease and is usually associated with hematological abnormality , including thrombocytopenia, the prevalence of which in SLE\patients has been reported to be 7-30%. Conversely, the prevalence of SLE in all ITP cases in adults is approximately 5%, making SLE the most common cause of secondary ITP. In the early stages, when there are only thrombocytopenia symptoms, it is sometimes difficult to determine what form of ITP is present in patients with SLE. SLE-associated thrombocytopenia (SLE- TP) is defined as a platelet count less than 100×109/L in the absence of any other identifiable cause.

The pathogenesis of thrombocytopenia in SLE is heterogeneous and multifactorial. However, it is widely accepted that an increased platelet clearance mediated by autoantibodies against platelets contributes to the pathogenesis, which is analogous to the mechanism of ITP. Differing from primary ITP, the clinical treatment for thrombocytopenia secondary to an identifiable cause is often targeted to the ongoing disorder. However, there are no specific biomarkers to differentiate SLE-TP from ITP.

The family of interleukin (IL)-1 cytokines is a family of protein molecules consisting of 11 members, including IL-1α (IL-1F1), IL-1β (IL-1F2), IL-1 receptor antagonist (IL-1Ra, IL-1F3), IL-18 (IL-1F4), IL-36Ra (IL-1F5), IL- 36α (IL-1F6), IL-37 (IL-1F7), IL-36β (IL-1F8), IL-36γ (IL-1F9), IL-38 (IL-1F10), and IL-33 (IL-1F11).

This cytokine family plays a crucial role as major proinflammatory and immunoregulatory mediators in a wide range of autoinflammatory, infectious, tumor, and autoimmune diseases that act through the receptors of the Toll-like/IL-1 receptor superfamily. The production of inflammatory cytokines such as IL-1, IL- 18, and IL-36 acts by activating target cells through the receptor superfamily then amplifying the immune response.

However, antagonists such as IL-1Ra, the receptor antagonist of IL-1α and IL-1β, act as inhibitors of IL-1 dependent inflammation. The blocking of IL-1, particularly of IL-1β, has recently become the standard therapy for autoinflammatory diseases. Moreover, IL-1β, a driver of tumor-promoting inflammation in cancer, can be targeted in patients using an IL-1 receptor antagonist acting as a checkpoint inhibitor. Several studies have suggested abnormal changes in IL-18, and IL-18-binding protein (IL-18BP) were involved in the pathogenesis of SLE and ITP .

Furthermore, recent studies demonstrate that IL-1 may also take part in inflammatory pathologies and auto-immune diseases by participating in the development of T-helper 17 (Th17) cells and increased numbers of Th17 cells have been reported in patients with SLE and ITP.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (18-60 years).

  * Diagnosed primary ITP
  * Diagnosed SLE with thrombocytopenia

Exclusion Criteria:

* • Patients on recent immunosuppressive therapy (<4 weeks).

  * Co-existing infections, malignancies, or other autoimmune cytopenias

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: It's a cross sectional study that will be carried out in the period from November 2025 to November 2026.
  * Groups:
    1. Group A: Patients with newly diagnosed or chronic primary ITP.
    2. Group B: Patients with SLE-associated thrombocytopenia.
    3. Group C: Healthy controls (age- and sex-matched).
       Inclusion Criteria:
  * Adults (18-60 years).
  * Diagnosed primary ITP
  * Diagnosed SLE with thrombocytopenia
  Exclusion Criteria:
  * Patients on recent immunosuppressive therapy (<4 weeks).
  * Co-existing infections, malignancies, or other autoimmune cytopenias.
  All patients will be subjected to : Sample Collection:
  * 5 ml peripheral blood collected under sterile conditions.
  * Separation of PBMCs (peripheral blood mononuclear cells).
  Laboratory Methods:
  1. RNA Extraction: from PBMCs.
  2. cDNA Synthesis: using reverse transcriptase.
  3. Gene Expression Analysis: using Quantitative Real-Time PCR (qRT-PCR)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1. To evaluate and compare the expression levels of IL-1β and IL-33 in patients with primary ITP and those with SLE-associated thrombocytopenia | January 2026 to August 2026
  * 5 ml peripheral blood collected under sterile conditions.
  * Separation of PBMCs (peripheral blood mononuclear cells).
  Laboratory Methods:
  1. RNA Extraction: from PBMCs.
  2. cDNA Synthesis: using reverse transcriptase.
  3. Gene Expression Analysis:
     * Quantitative Real-Time PCR (qRT-PCR)
2. To correlate cytokine expression levels with platelet counts and disease activity scores. | January 2026 to August 2026
  * 5 ml peripheral blood collected under sterile conditions.
  * Separation of PBMCs (peripheral blood mononuclear cells).
  Laboratory Methods:
  1. RNA Extraction: from PBMCs.
  2. cDNA Synthesis: using reverse transcriptase.
  3. Gene Expression Analysis:
     * Quantitative Real-Time PCR (qRT-PCR)
3. To assess the potential of IL-1β and IL-33 as diagnostic biomarkers for differentiating ITP from SLE-thrombocytopenia. | June 2026 to august 2026
  * 5 ml peripheral blood collected under sterile conditions.
  * Separation of PBMCs (peripheral blood mononuclear cells).
  Laboratory Methods:
  1. RNA Extraction: from PBMCs.
  2. cDNA Synthesis: using reverse transcriptase.
  3. Gene Expression Analysis:
     * Quantitative Real-Time PCR (qRT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Z elsayed, Lecturer, Principal Investigator — faculty of Medicine Sohag university; Samar M Kamal, lecturer, Study Chair — fauculty of Medicine , Sohag university

IPD SHARING:
Plan to Share IPD: No